CLINICAL TRIAL: NCT02313246
Title: A Pilot Study of Cognitive-Behaviour Therapy for Irritable Bowel Syndrome and the Gut Microbiome
Acronym: IBS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left the institution
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBT-IBS-2015
Record Dates: First submitted 2014-12-05; First posted 2014-12-10 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group Cognitive Behaviour Therapy (Experimental): Patients will complete an 11-session group cognitive behaviour therapy for IBS that will be led by two clinicians, one of whom will be a registered clinical psychologist, at the Digestive Diseases Clinic at McMaster University Medical Centre. The group cognitive behaviour therapy will include weekly 2-hour sessions for 11 weeks. Sessions will cover the following topics: psychoeducation about IBS and the role of stress in exacerbating IBS symptoms, progressive muscle relaxation, stress management, problem solving, identifying and modifying maladaptive thinking patterns, decreasing behavioural avoidance, and exposure to feared physical sensations.
  Interventions: Behavioral: Group Cognitive Behaviour Therapy

INTERVENTIONS:
Behavioral: Group Cognitive Behaviour Therapy — This 11-week group treatment will cover the following topics: psychoeducation about IBS and the role of stress in exacerbating IBS symptoms, progressive muscle relaxation, stress management, problem solving, identifying and modifying maladaptive thinking patterns, decreasing behavioural avoidance, and exposure to feared physical sensations.

SUMMARY:
This study evaluates the effectiveness of a group cognitive behaviour therapy for Irritable Bowel Syndrome (IBS) in decreasing symptoms of IBS, improving quality of life, and normalizing the gut microbiome. Patients will complete an 11-week group cognitive behaviour therapy for IBS within 1 month of being deemed eligible for the study.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a chronic, disabling functional gastrointestinal disorder that is characterized by abdominal pain or discomfort and a disturbance in bowel habit. Approximately five million Canadians currently suffer with this chronic illness, which can have a significant impact on work and school absenteeism, productivity, social functioning and quality of life (Fedorak et al., 2012). Although the etiology of IBS is still unclear, there is increased interest in the role of the gut-brain axis in the development and maintenance of IBS. A growing body of evidence has identified changes in the composition, temporal stability and metabolic activity of the gut microbiome in IBS (Bolino & Bercik, 2010). Moreover, there is evidence for bidirectional communication between the gut and the brain, such that the gut microbiota appear to influence as well as be modulated by brain activity through neurohumoral mechanisms (Collins, Surette, & Bercik, 2012).

Currently, medications are the most widely used treatment for IBS (Ford et al., 2009; Ford et al., 2014). Although there is good evidence for the effectiveness of medications in reducing IBS symptomatology and improving quality of life, these medications are also often associated with unpleasant side effects. As a result, there is a growing interest in the utilization of psychological treatments, including cognitive behaviour therapy, for IBS. Cognitive behaviour therapy is a psychotherapeutic approach that addresses maladaptive cognitive processes and behaviours in a systematic, explicit fashion. Although there is good evidence for the effectiveness of cognitive behaviour therapy for the treatment of IBS (Ford et al., 2009; Ford et al., 2014), there is a lack of research examining the mechanisms through which cognitive behaviour therapy influences symptoms of IBS.

Accordingly, the current study has three aims: 1) to evaluate the effectiveness of group cognitive behaviour therapy for IBS on IBS symptomatology and quality of life; 2) to examine whether there are any changes in the gut microbiome from pre to posttreatment; and 3) to examine whether changes in the gut microbiome following cognitive behaviour therapy mediate changes in IBS symptomatology and quality of life. The current study has the potential of increasing knowledge about the role of the gut microbiome in IBS as well as the mechanisms of cognitive behaviour therapy for IBS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with irritable bowel syndrome
* Able to commit to attending weekly 2-hour group sessions for 12 weeks

Exclusion Criteria:

* Use of antibiotics, or probiotics during the 4-week period prior to enrolling in the study
* Changes in medications during the 4-week period prior to enrolling in the study
* Presence of a major medical illness that may change the gut microbiome (e.g., any comorbid gastroenterological, rheumatological, or immunological disorder)
* Diagnosis of a major psychiatric disorder that is likely to impede participation in group therapy (e.g., depression with active suicidality, psychosis, or gross cognitive impairment)
* Received psychotherapy for IBS within the past 5 years
* Inability to read or complete symptom diaries or questionnaires
* Inability or unwillingness to provide or sign informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Birmingham IBS Symptom Scale | baseline to 11 weeks
IBS Quality of Life | Baseline to 11 weeks
Changes in gut microbiome as assessed through analyzing fecal samples | Baseline to 6 weeks
Changes in gut microbiome as assessed through analyzing fecal samples | Baseline to 11 weeks

SECONDARY OUTCOMES:
GI-Cognitions Questionnaire | Baseline to 6 weeks
GI-Cognitions Questionnaire | Baseline to 11 weeks
Visceral Sensitivity Index | Baseline to 6 weeks
Visceral Sensitivity Index | Baseline to 11 weeks
Visceral Sensitivity Index | 11 weeks to 15 weeks
Hospital Anxiety and Depression Scale | Baseline to 6 weeks
Hospital Anxiety and Depression Scale | Baseline to 11 weeks
Penn State Worry Questionnaire | Baseline to 6 weeks
Penn State Worry Questionnaire | Baseline to 11 weeks
UCLA Symptom Severity Scale | Weekly for 11 weeks
UCLA Symptom Severity Scale | 11 weeks to 15 weeks
Irritable Bowel Syndrome Symptom Severity Scale | Weekly for 11 weeks
Anxiety Sensitivity Index | Baseline to 6 weeks
Anxiety Sensitivity Index | Baseline to 11 weeks
IBS Quality of Life | 11 weeks to 15 weeks
Birmingham IBS Severity Scale | 11 weeks to 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matilda E. Nowakowski, PhD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fedorak RN, Vanner SJ, Paterson WG, Bridges RJ. Canadian Digestive Health Foundation Public Impact Series 3: irritable bowel syndrome in Canada. Incidence, prevalence, and direct and indirect economic impact. Can J Gastroenterol. 2012 May;26(5):252-6. doi: 10.1155/2012/861478. PMID 22590697
- [Result] Ford AC, Talley NJ, Schoenfeld PS, Quigley EM, Moayyedi P. Efficacy of antidepressants and psychological therapies in irritable bowel syndrome: systematic review and meta-analysis. Gut. 2009 Mar;58(3):367-78. doi: 10.1136/gut.2008.163162. Epub 2008 Nov 10. PMID 19001059
- [Result] Ford AC, Quigley EM, Lacy BE, Lembo AJ, Saito YA, Schiller LR, Soffer EE, Spiegel BM, Moayyedi P. Effect of antidepressants and psychological therapies, including hypnotherapy, in irritable bowel syndrome: systematic review and meta-analysis. Am J Gastroenterol. 2014 Sep;109(9):1350-65; quiz 1366. doi: 10.1038/ajg.2014.148. Epub 2014 Jun 17. PMID 24935275
- [Result] Collins SM, Surette M, Bercik P. The interplay between the intestinal microbiota and the brain. Nat Rev Microbiol. 2012 Nov;10(11):735-42. doi: 10.1038/nrmicro2876. Epub 2012 Sep 24. PMID 23000955
- [Result] Bolino CM, Bercik P. Pathogenic factors involved in the development of irritable bowel syndrome: focus on a microbial role. Infect Dis Clin North Am. 2010 Dec;24(4):961-75, ix. doi: 10.1016/j.idc.2010.07.005. PMID 20937460